CLINICAL TRIAL: NCT00981175
Title: Randomised, Double-blind, Phase 2 Study of the Safety, Immunogenicity and Duration of Immunity of ChimeriVax™-JE, Live Attenuated Vaccine in Healthy Adults
Brief Title: A Study of ChimeriVax™-JE Live Attenuated Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-005
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Encephalitis; Japanese Encephalitis
Keywords: Japanese Encephalitis; Japanese Encephalitis Vaccines; Adult
MeSH Terms: conditions — Encephalitis; Encephalitis, Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group 1: ChimeriVax™-JE Vaccine first, then Placebo (Experimental): Participants received ChimeriVax™-JE on Day 0 and ChimeriVax diluent on Day 28
  Interventions: Biological: Live attenuated Japanese encephalitis virus, then ChimeriVax diluent
- Study Group 2: Placebo first, then ChimeriVax™-JE Vaccine (Experimental): Participants received ChimeriVax diluent on Day 0 and ChimeriVax™-JE on Day 28.
  Interventions: Biological: ChimeriVax diluent, then Live attenuated Japanese encephalitis virus

INTERVENTIONS:
Biological: Live attenuated Japanese encephalitis virus, then ChimeriVax diluent — ChimeriVax™-JE, 0.5 mL subcutaneous on Day 0; ChimeriVax diluent 0.5 mL subcutaneous on Day 28
  Other Names: ChimeriVax™-JE
  Arms: Study Group 1: ChimeriVax™-JE Vaccine first, then Placebo
Biological: ChimeriVax diluent, then Live attenuated Japanese encephalitis virus — ChimeriVax diluent, 0.5 mL subcutaneous on Day 0 and ChimeriVax™-JE, 0.5 mL subcutaneous on Day 28.
  Other Names: ChimeriVax™-JE
  Arms: Study Group 2: Placebo first, then ChimeriVax™-JE Vaccine

SUMMARY:
The purpose of this study is to assess the safety, tolerability, immunogenicity, and duration of immunity of one or two doses of ChimeriVax™-JE vaccine separated by 5 or 6 months in adults.

Objectives:

Safety:

* Obtain safety and tolerability data of a single, fixed dose of ChimeriVax™-JE compared with a placebo in adult volunteers (≥ 18 to <55 years) without prior Japanese encephalitis (JE) vaccination.

Immunogenicity:

* Obtain data on the antibody response in adult volunteers following administration of ChimeriVax™-JE
* Assess the durability of the immune response in adult volunteers over 60 months following one or two doses of ChimeriVax™-JE.

DETAILED DESCRIPTION:
Participants will receive ChimeriVax™-JE or diluent on Day 0 and diluent or ChimeriVax™-JE on Day 28. A subset of participants in each group will receive a booster dose of ChimeriVax™-JE at Month 6. Follow-up visits will occur at 12 and 24 months. Eligible participants will then enter the long-term immunogenicity follow-up period with visits at approximately 36, 48, and 60 months after Day 0. No safety data will be collected in the long-term immunogenicity follow-up period.

ELIGIBILITY:
Inclusion Criteria :

At entry:

* All aspects of the protocol explained and written informed consent obtained from the subject.
* Aged ≥ 18 to < 55 years.
* In good general health, without significant medical history, physical examination findings, or clinically significant abnormal laboratory results.
* Subject must be available for the study duration, including all planned follow-up visits.
* Has the subject agreed to take the following precautions to avoid insect bites for 7 days following vaccination: (a) wear long-sleeved shirts and trousers?; (b) apply N,N-Diethyl-meta-toluamide (DEET)-containing insect repellents?; (c) Sleep in screened enclosures?
* For female subjects of childbearing potential: Negative serum pregnancy tests. An efficacious hormonal (i.e., oral, implantable or injectable) or barrier method of birth control must be used at least 1 month before Screening and Month 6 and at least 1 month after Day 28 and Month 6. These subjects will sign an agreement that birth control will be practised during the specified periods and will specify the method used. Female subjects unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).

For long-term immunogenicity follow-up period:

* Subject received an initial dose of ChimeriVax™-JE, has a baseline (Day 0) sample and at least one post-vaccination evaluable serological specimen for antibody analysis.
* All aspects of the Long-term Immunogenicity Follow-up Period explained and updated written informed consent obtained from the subject.
* In good general health, without significant medical history that may affect the efficacy endpoints or the ability to take blood samples.

Exclusion Criteria :

* A history of vaccination to Japanese encephalitis (JE). Previous vaccination will be determined by history (interview of subject) and/or by reviewing the subject's vaccination card or other official documentation (either a history of or documentation of vaccination fulfils the criterion for exclusion).
* Known or suspected immunodeficiency (e.g., human immunodeficiency virus [HIV] infection, primary immunodeficiency disorder, leukemia, lymphoma), use of immunosuppressive or antineoplastic drugs (corticosteroids > 10 mg prednisone, or equivalent, for more than 14 days in the last three months).
* Clinically significant abnormalities on laboratory assessment.
* Serious adverse reactions characterised by urticaria or angioedema to a prior vaccine.
* Transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within six months of the Screening Visit or up to Day 56.
* Administration of another vaccine within 30 days preceding the screening visit or up to Day 56 (these subjects will be rescheduled for vaccination at a later date).
* Physical examination indicating any clinically significant medical condition.
* Body temperature >38.1°C (100.6°F) or acute illness within 3 days prior to inoculation (subject may be rescheduled).
* Intention to travel out of the area prior to the study visit on Day 56.
* Seropositive to hepatitis C virus (HCV) or HIV or positive for hepatitis B (HBV) (antigen).
* Lactation or intended pregnancy in female subjects.
* Excessive alcohol consumption, drug abuse, significant psychiatric illness.
* A known or suspected physiological or structural condition that compromises the integrity of the blood-brain barrier (e.g., significant hypertensive cerebrovascular disease, trauma, ischemia, infection, inflammation of the brain).

For long-term immunogenicity follow-up period:

* History of Yellow Fever or out of study JE vaccination or known flavivirus infection since receiving ChimeriVax™-JE vaccination on Day 0 or Day 28 (during double-blind treatment period of the study). Yellow Fever/JE vaccination or flavivirus infection will be determined by history (interview of subject) and/or by reviewing the subject's medical records. Please note subjects who were flavivirus positive at Day 0 will be allowed to enrol on the study.
* Participation in another JE clinical study.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2003-04; Primary Completion 2004-06 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Enoggera, Queensland, Australia

REFERENCES:
- [Result] Nasveld PE, Ebringer A, Elmes N, Bennett S, Yoksan S, Aaskov J, McCarthy K, Kanesa-thasan N, Meric C, Reid M. Long term immunity to live attenuated Japanese encephalitis chimeric virus vaccine: randomized, double-blind, 5-year phase II study in healthy adults. Hum Vaccin. 2010 Dec;6(12):1038-46. doi: 10.4161/hv.6.12.13057. Epub 2010 Dec 1. PMID 21150279
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and vaccinated from 14 April 2003 to 05 January 2004 at 1 clinical center in Australia.
Pre-assignment Details: A total of 202 participants who met the inclusion/exclusion criteria were enrolled and vaccinated. A subset of the participants also received a booster vaccine at month 6. A report on all participants who received the primary and booster vaccination and the primary vaccination only are presented.
Groups:
- ChimeriVax™-JE Vaccine First, Then Placebo: Participants received ChimeriVax™-JE vaccine on Day 0 and vaccine diluent (placebo) on day 28.
- Placebo First, Then ChimeriVax™-JE Vaccine: Participants received vaccine diluent (placebo) on Day 0 and ChimeriVax™-JE vaccine on day 28.
Period: Primary Dose Vaccination
Arm/Group | ChimeriVax™-JE Vaccine First, Then Placebo | Placebo First, Then ChimeriVax™-JE Vaccine
Started | 101 | 101
Completed | 98 | 99
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Period: Booster Dose Vaccination
Arm/Group | ChimeriVax™-JE Vaccine First, Then Placebo | Placebo First, Then ChimeriVax™-JE Vaccine
Started | 55 (A sub-set of participants in the group received the booster ChimeriVax™-JE vaccine.) | 43 (A sub-set of participants in the group received the booster ChimeriVax™-JE vaccine.)
Completed | 53 | 40
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- ChimeriVax™-JE Vaccine First , Then Placebo: Participants received ChimeriVax™-JE vaccine on Day 0 and vaccine diluent (placebo) on Day 28.
- Booster ChimeriVax™-JE Vaccine: Participants received a booster dose of ChimeriVax™-JE vaccine at Month 6 Following vaccination with ChimeriVax™-JE vaccine and Diluent (Placebo) at Day 0 and Day 28
- Total: Total of all reporting groups
Arm/Group | ChimeriVax™-JE Vaccine First , Then Placebo | Placebo First, Then ChimeriVax™-JE Vaccine | Booster ChimeriVax™-JE Vaccine | Total
Number analyzed (Participants) | 101 | 101 | 0 | 202
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 101 | 101 |  | 202
  >=65 years | 0 | 0 |  | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 26.1 (7.36) | 27.7 (8.25) |  | 26.9 (7.84)
Gender [Number; unit: participants]
  Female | 13 | 15 |  | 28
  Male | 88 | 86 |  | 174
Region of Enrollment [Number; unit: participants]
  Australia | 101 | 101 |  | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seroconversion to Homologous ChimeriVax-JE Virus Strain After a Single Dose of Chimerivax™-JE and Placebo Dose
Description: Assay by 50% Plaque Reduction Neutralization Test (PRNT50) Seroconversion: PRNT50 ≥ 10 and PRNT50 ≥ 20. Assessed in all participants who received ChimeriVax™-JE vaccine on Day 0 and Day 28.
Time Frame: Day 28 post-vaccination
Population: Immunogenicity was assessed in the Intent-to-Treat Population.
Measure: Number; unit: Participants
Groups:
- ChimeriVax™-JE Vaccine (Single or Primary): Outcome for all participants that received ChimeriVax™-JE vaccine on Day 0 or day 28.
- Booster ChimeriVax™-JE Vaccine: Participants received ChimeriVax™-JE vaccine booster at month 6.
- No Booster Vaccine: Participants did not receive a booster dose Chimerivax™-JE vaccine
Arm/Group | ChimeriVax™-JE Vaccine (Single or Primary) | Booster ChimeriVax™-JE Vaccine | No Booster Vaccine
Number analyzed (Participants) | 201 | 0 | 0
Participants
  PRNT50 ≥ 10 [N = 197] | 194 |  |
  PRNT50 ≥ 20 [N = 197] | 191 |  |

2. Secondary Outcome: Number of Participants With Seroconversion to Homologous ChimeriVax™-JE Virus Strain After a Single Dose of Chimerivax™-JE and Placebo Followed by a Booster Vaccine Dose.
Description: Assay by 50% Plaque Reduction Neutralization Test (PRNT50) Seroconversion: PRNT50 ≥ 10 and PRNT50 ≥ 20. Assessed in all participants who received ChimeriVax™-JE vaccine on Day 0 and Day 28 and pre- and post-Booster vaccination.
Time Frame: Month 6 pre- and post-vaccination
Population: Immunogenicity was assessed in the Intent to Treat Population pre- and post-booster vaccination.
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE Vaccine (Single or Primary) | Booster ChimeriVax™-JE Vaccine | No Booster Vaccine
Number analyzed (Participants) | 0 | 97 | 103
Participants
  Pre-booster PRNT50 ≥ 10 [N = 0, 98, 93] |  | 95 | 90
  Post-booster PRNT50 ≥ 10 [N = 0, 97, 0] |  | 97 | NA — Participants did not receive treatment
  Pre-booster PRNT50 ≥ 20 [N = 0, 98, 93] |  | 93 | 87
  Post-booster PRNT50 ≥ 20 [N = 0, 97, 0] |  | 97 | NA — Participants did not receive treatment

3. Secondary Outcome: Number of Participants With Seroconversion to Homologous ChimeriVax™-JE Virus Strain After a Single Dose of Chimerivax™-JE and Placebo Followed or Not by a Booster Vaccine Dose at 6 Month.
Description: Assay by 50% Plaque Reduction Neutralization Test (PRNT50) Seroconversion: PRNT50 ≥ 10 and PRNT50 ≥ 20. Assessed in all participants who received ChimeriVax™-JE vaccine on Day 0 and Day 28 and followed or not by a booster vaccine dose at 6 month.
Time Frame: Month 12 post-vaccination
Population: Immunogenicity was assessed in the Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE Vaccine (Single or Primary) | Booster ChimeriVax™-JE Vaccine | No Booster Vaccine
Number analyzed (Participants) | 0 | 97 | 103
Participants
  PRNT50 ≥ 10 [N = 0, 80, 76] |  | 79 | 72
  PRNT50 ≥ 20 [N = 0, 80, 76] |  | 78 | 68

4. Secondary Outcome: Number of Participants With Seroconversion to Homologous ChimeriVax-JE Virus Strain After a Single Dose of Chimerivax™-JE and Placebo Followed or Not by a Booster Vaccine Dose at 6 Month.
Description: Assay by 50% Plaque Reduction Neutralization Test (PRNT50) Seroconversion: PRNT50 ≥ 10 and PRNT50 ≥ 20. Assessed in all participants who received ChimeriVax™-JE vaccine on Day 0 and Day 28 and followed or not by a booster vaccine dose at month 24.
Time Frame: Month 24 post-vaccination
Population: Immunogenicity was assessed in the Intent to Treat Population
Measure: Number; unit: Participants
Arm/Group | ChimeriVax™-JE Vaccine (Single or Primary) | Booster ChimeriVax™-JE Vaccine | No Booster Vaccine
Number analyzed (Participants) | 0 | 97 | 103
Participants
  PRNT50 ≥ 10 [N = 0, 70, 71] |  | 69 | 64
  PRNT50 ≥ 20 [N = 0, 70, 71] |  | 67 | 60

5. Primary Outcome: Number of Participants Reporting Injection Site Treatment Emergent Adverse Events Post-Vaccination With ChimeriVax™-JE or Placebo at Day 0 and Day 28, and Following a Booster of ChimeriVax™-JE at Month 6 in a Subset of the Study Population.
Description: Injection Site Treatment Emergent Adverse Events: Pain, Reaction Not Otherwise Specified (NOS), Erythema, Swelling, Bruising, Nodule, Pigmentation Changes, Pruritus were assessed in all participants for up to 28 days post-Vaccination.
Time Frame: Days 0 to 28 post-vaccination
Population: Injection site reactions were assessed in the Safety Population.
Measure: Number; unit: Participants
Groups:
- ChimeriVax™-JE Vaccine: Participants received a primary dose of ChimeriVax™-JE vaccine at either Day 0 or Day 28
- Placebo Vaccine: Participants received a dose of placebo vaccine (diluent)at either Day 0 or Day 28
Arm/Group | ChimeriVax™-JE Vaccine | Placebo Vaccine | Booster ChimeriVax™-JE Vaccine
Number analyzed (Participants) | 201 | 199 | 98
Participants
  Injection site Pain | 7 | 5 | 0
  Injection site Reaction NOS | 6 | 4 | 0
  Injection site Erythema | 4 | 5 | 0
  Injection site Swelling | 2 | 6 | 1
  Injection site Bruising | 1 | 1 | 0
  Injection site Nodule | 1 | 0 | 0
  Injection site Pigmentation Changes | 1 | 1 | 0
  Injection site Pruritus | 1 | 0 | 0

6. Secondary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events Recorded as Possibly, Probably, or Definitely Related to Study Treatment.
Description: Treatment emergent adverse events were assessed in all participants receiving ChimeriVax-JE Vaccine, Diluent (Placebo), or Booster Vaccination.
Time Frame: Day 0 up to 28 post-vaccination
Population: Treatment emergent adverse events were assessed in the Safety Population.
Measure: Number; unit: Participants
Groups:
- Placebo Vaccine: Participants received a dose of placebo vaccine (diluent) at either Day 0 or Day 28
- Booster ChimeriVax™-JE Vaccine: Participants received a booster dose of ChimeriVax™-JE vaccine at month 6 following primary ChimeriVax™-JE and Diluent vaccination at Day 0 and Day 28
Arm/Group | ChimeriVax™-JE Vaccine | Placebo Vaccine | Booster ChimeriVax™-JE Vaccine
Number analyzed (Participants) | 201 | 199 | 98
Participants
  Any Adverse Event | 47 | 45 | 4
  Headache | 12 | 10 | 0
  Injection Site Pain | 7 | 5 | 0
  Injection Site Reaction Not Otherwise Specified | 6 | 4 | 0
  Lethargy | 5 | 2 | 0
  Viral Infection Not Otherwise Specified | 5 | 10 | 0
  Injection Site Erythema | 4 | 5 | 0
  Fatigue | 3 | 2 | 0
  Lymphadenopathy | 2 | 0 | 0
  Injection Site Swelling | 2 | 6 | 1
  Diarrhea Not Otherwise Specified | 2 | 1 | 0
  Nausea | 2 | 2 | 0
  Pyrexia | 2 | 2 | 3
  Liver Function Test Abnormal | 2 | 2 | 0
  Myalgia | 2 | 2 | 0
  Upper Respiratory Tract Infection NOS | 2 | 9 | 0
  Vomiting Not Otherwise Specified | 1 | 0 | 0
  Injection Site Bruising | 1 | 1 | 0
  Injection Site Nodule | 1 | 0 | 0
  Injection Site Pigmentation Changes | 1 | 1 | 0
  Injection Site Pruritus | 1 | 0 | 0
  Malaise | 1 | 2 | 0
  Rigors | 1 | 0 | 0
  Gastroenteritis Not Otherwise Specified | 1 | 0 | 0
  Anorexia | 1 | 0 | 0
  Pharygolaryngeal Pain | 1 | 0 | 0
  Insomnia | 0 | 1 | 0
  Dry Eyes Not Otherwise Specified | 0 | 1 | 0
  Disturbance in Attention | 0 | 1 | 0
  Contusion | 0 | 1 | 0
  Flushing | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from day of vaccination (Day 0) for up to 6 months post-vaccination.
Arm/Group | ChimeriVax™-JE Vaccine First , Then Placebo | Placebo First, Then ChimeriVax™-JE Vaccine | Booster ChimeriVax™-JE Vaccine
Serious Adverse Events (participants affected / at risk) | 2/201 | 1/199 | 0/98
Other Adverse Events (participants affected / at risk) | 27/201 | 35/199 | 3/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChimeriVax™-JE Vaccine First , Then Placebo (N=201) | Placebo First, Then ChimeriVax™-JE Vaccine (N=199) | Booster ChimeriVax™-JE Vaccine (N=98)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Not Otherwise Specified (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Infection Not Otherwise Specified (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChimeriVax™-JE Vaccine First , Then Placebo (N=201) | Placebo First, Then ChimeriVax™-JE Vaccine (N=199) | Booster ChimeriVax™-JE Vaccine (N=98)
Diarrhea Not Otherwise Specified (Gastrointestinal disorders) | 2 (2) | 6 (6) | 1 (1)
Injection Site Pain (General disorders) | 7 (7) | 5 (5) | 0 (0)
Injection Site Reaction Not Otherwise Specified (General disorders) | 6 (6) | 4 (4) | 0 (0)
Injection Site Swelling (General disorders) | 2 (2) | 6 (6) | 1 (1)
Lethargy (General disorders) | 11 (11) | 5 (5) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 3 (3)
Upper Respiratory Tract Infection NOS (Infections and infestations) | 24 (27) | 35 (38) | 1 (1)
Viral Infection Not Otherwise Specified (Infections and infestations) | 5 (5) | 11 (11) | 0 (0)
Headache (Nervous system disorders) | 27 (31) | 20 (20) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications